CLINICAL TRIAL: NCT02155569
Title: Extraperitoneal Versus Transperitoneal Cesarean Section: A Prospective Randomized Comparison
Brief Title: Extraperitoneal Versus Transperitoneal Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ragıp Atakan Al, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: atauni8
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Cesarean, Extraperitoneal
Keywords: Cesarean, extraperitoneal; Cesarean; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transperitoneal Cesarean (Active Comparator)
  Interventions: Procedure: Transperitoneal Cesarean
- Extraperitoneal Cesarean (Active Comparator)
  Interventions: Procedure: Extraperitoneal Cesarean

INTERVENTIONS:
Procedure: Extraperitoneal Cesarean — Pfannenstiel incision, paravesical approach to lower uterine segment extraperitoneally and Kerr incision for uterine entry
  Arms: Extraperitoneal Cesarean
Procedure: Transperitoneal Cesarean — Pfannenstiel-Kerr technique for laparatomy and uterine entry
  Arms: Transperitoneal Cesarean

SUMMARY:
The aim of the study is to compare post operative morbidity between extra peritoneal cesarian and trans peritoneal cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean (primary or repeated up to four)

Exclusion Criteria:

* emergent cesarean
* macrosomia (fetal weight > 4500 g)
* history of major abdominal surgery
* suspected abnormal placentation
* placenta previa

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
post operative pain | One hour before cesarean and 24 hour postoperatively
  Perceived pain scores will be measured by an visual analog scale.

SECONDARY OUTCOMES:
delivery time | 2 minutes after delivery
  skin incision to delivery
operation time | 5 minutes postoperatively
  skin incision to skin closure
hemoglobin differences | one hour before cesarean, 48 hour postoperatively
need for extra analgesic | 48 hour
nausea | 48 hour
vomiting | 48 hour
thoracic and shoulder pain | 48 hour
Urogenital distress measured by Urogenital Distress Inventory | One hour before cesarean and 24 hour postoperatively
Oral intake | 48 hour
  The percentage of patients who tolerates oral intake. Oral intake will be allowed 4-6 hour after cesarean for extraperitoneal group. For intraperitoneal group it will be allowed when patient passed gas.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)